CLINICAL TRIAL: NCT05071417
Title: Effect Of Semaglutide In Coronary Atherosclerotic Plaqus Assessed by Coronay CT
Brief Title: Effect Of Semaglutide In Coronary Atheroma Plaque
Acronym: SEPLA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Responsible Party: Principal Investigator, PM1-SEPLA IBSAL, Professor, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEPLA
Record Dates: First submitted 2021-08-05; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Atheroscleroses, Coronary
MeSH Terms: conditions — Coronary Artery Disease | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Phase IV low-intervention, double-blind, multicenter clinical trial to evaluate the effects of 18 months of semaglutide treatment on the volume, architecture, and composition of coronary atheroma plaques in subjects with DM2 for at least 10 years and without clinical cardiovascular disease.
  Patients with DM2 will be included if their previously prescribed treatment was insufficient to achieve adequate control of glycemic and glycosylated hemoglobin levels (HBA1c) to reach their therapeutic objective and the researcher has considered semaglutide treatment to be appropriate according to its clinical criteria and based on the indication of this treatment in this patient profile. The study treatment will therefore be the same treatment that the patient would receive even if they did not participate in the study; this condition is the basic norm for the inclusion of the patient in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Experimental): Patients on semaglutide
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Usual treatment with semaglutide. Dose 0.5 - 1mg weekly, subcutaneous, weekly

SUMMARY:
The main objective of this trial is to evaluate the effect of Semaglutide on the burden of coronary atherosclerosis, based on the change in Percent Atheroma Volume (PAV) by quantifying atheroma plaque throughout the coronary tree based on the analysis of CCTA in asymptomatic subjects with T2D in optimized and stable treatment with Semaglutide.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (DM2) are considered to be at high vascular risk (VR). However, the VR risk may vary, depending on the presence of other cardiovascular risk factors (CVRFs), particularly dyslipidemia, smoking habit, hypertension, and obesity. High blood glucose levels are part of the etiopathogenic basis of atherosclerosis, whose vascular complications are the leading cause of death and disability in developed countries. Atherosclerosis is considered a chronic immunoinflammatory process with a polygenic and multifactorial origin that begins early due to vascular endothelial dysfunction. Atherosclerosis is a dynamic process that develops intermittently over time; periods of inactivity and rapid evolution are interspersed and modulated by environmental and genetic factors. As a result of a series of etiopathogenic and environmental factors, lesions (plaques) develop with greater or lesser lipid content, collagen, elastic fibers, and calcium. The location and degree of development of atherosclerotic plaques give rise to different forms of atherosclerotic disease, which is characterized by symptoms and signs that correspond to the obstruction of the vascular lumen with decreased flow and the consequent occurrence of (possibly chronic) ischemia. Atherosclerotic disease can also be characterized by the rupture of the plaque and the appearance of thrombotic phenomena (because the lipid nucleus of the plaque is highly thrombogenic and triggers the activation of the coagulation and platelet adhesion and aggregation cascades), with manifestations of acute ischemia.

The relationship between the composition of the atheroma plaque and the occurrence of cardiovascular events, revealed the need for imaging techniques that could identify not only the degree of stenosis of atherosclerotic lesions, but also their volume, composition and levels of inflammation, and thus being able to identify the possible high-risk plaques (vulnerable plaques). Within imaging techniques, there are invasive ones such as coronary angiography or coronary angiography, ultrasound or intravascular ultrasound (IVUS) and optical coherence tomography (OCT); and non-invasive, such as magnetic resonance imaging (MRI), positron emission tomography (PET), and computed tomography.

Invasive coronary angiography has traditionally been the reference imaging test to determine the degree of stenosis and continues to be the procedure of choice for the evaluation of coronary anatomy and the identification of atherosclerotic lesions. Angiography provides information on the number and size of vascular stenosis but does not allow to know the plaque composition. Provides Simply an image of the internal arterial lumen but lacks the ability to adequately represent the vessel wall with its developing atherosclerotic plaque.

Intravascular ultrasound (IVUS) is considered the reference method for the evaluation of atherosclerotic plaque burden and plaque characteristics. However, IVUS is an invasive method that has risks, cannot be used to study the entire coronary tree, only in one segment of the arterial tree and is not indicated for asymptomatic individuals.

The IVUS technique plus virtual histology allows the identification of atheroma plaques in the vascular tree, and can quantify the size, volume, composition and distribution of the plaque. However, a limitation of this technique is the ability of the ultrasound signal to penetrate the calcified tissue, resulting in an acoustic shadow after the calcified tissue.

Currently, with the new advances in the development of cardiac imaging techniques, coronary computed tomographic angiography (CCTA) has been incorporated as a non-invasive and easily applied method for direct visualization of coronary arteries without the need to introduce a catheter The image study of the coronary vessels by CCTA has been proposed as a suitable method for the qualitative detection of changes in the vessel wall, allowing the evaluation of the coronary arteries and the characterization of the atherosclerotic plaque.

In the last decade, several advances have been seen in CCTA that have made it one of the key diagnostic instruments for the non-invasive evaluation of coronary atherosclerosis in patients with a low to intermediate probability of coronary heart disease. CCTA may be useful for prognostic classification together with classic CVRF in patients with intermediate cardiovascular risk, for more accurate reclassification and as a screening for the early diagnosis of coronary atherosclerotic disease in certain groups of patients at special risk.

Previous studies have shown that CCTA is comparable to IVUS for the classification of atheroma plaques. CCTA, therefore, emerges as a non-invasive alternative for plaque characterization compared to other techniques such as IVUS.

Coronary CCTA has established itself as a reliable and accurate tool for the detection of coronary atherosclerotic plaque and stenosis. Since CCTA provides information about plaque burden and the characteristics of high-risk plaques, the addition of these parameters to the traditional interpretation of CCTA, which is limited to the detection of stenosis, could improve the efficiency of this method for the early detection of coronary heart disease.

Plaque characteristics are usually analyzed in a qualitative (subjective) way. This limitation can be solved through the use of new analytical platforms that allow automated quantification of the characteristics of the coronary plaque with high accuracy and reproducibility. In this context, software tools have been developed for the automated quantification of atheroma plaques in CCTA images. In this area, the QAngio CT (Medis medical imaging system, the netherlans) stands out, a software tool designed to perform quantitative analysis of images in CCTA data sets. In the CCTA data sets, the software is able to detect the contours of the vessel wall and the lumen, which are used for automated quantitative evaluations of coronary plaques. As for the characterization of the atherosclerotic plaque, the software is able to analyze virtual histology, differentiating between what is the mean, fibrous plaque, fibro-fatty, necrotic and calcified, with its consequent prognostic implication. The parameters of the entire coronary tree are obtained independently: vessel length, plaque burden, plaque volume, maximum thickness of the plaque, volume and percentage of fibrous plaque, fibro-fatty plaque, necrotic plaque and calcium plaque, maximum stenosis by area and by diameter. This software tool has a number of advantages over the analysis based on the IVUS. First, the non-invasiveness of the CCTA technique based on which this tool performs quantitative plaque analysis allows a consecutive analysis with a lower risk than that of IVUS. In addition, previous studies have demonstrated the correlation between QAngio CT and IVUS-based analysis regarding the area of lumen stenosis, plaque burden and remodeling index. On the other hand, although IVUS is the reference method for plaque quantification, it has the limitation of analyzing only a specific segment of the coronary tree, while QAngio CT allows the complete analysis of the coronary tree. In an evaluation study of atheroma plaque, this method could provide information not only on the size of the plaque, but also on the characteristics of the plaque.

The change in plaque volume has been used successfully to monitor plaque progression in studies with IVUS. Using IVUS, plaque volumes are calculated as the difference between the area of the outer elastic membrane and the lumen area for successive cross sections of a coronary artery. The difference between the volume of the vessel and the volume of the lumen constitutes the total volume of the plaque. From these volumes, other parameters such as the plaque burden or percentage of atheroma volume (PVA) or the total volume of atheroma (VTA) can be derived, being PVA the most reproducible and the molt related to cardiovascular prognosis.

Furthermore, recent studies have correlated the evaluation of the radiographic characteristics of plaque (Virtual histology) with the patient's prognosis. The QAngio CT provides an automated evaluation of the characteristics of the complete coronary tree plate based on radiological densities.

The prevention and treatment of DM2 should be considered an essential part of atherosclerotic disease. Throughout numerous and extensive clinical trials, it has been shown that reductions in blood glucose and HbA1c levels lead to reductions in cardiovascular risks. This knowledge suggests that atherosclerosis can be influenced by DM2 treatment.

Numerous studies have shown the beneficial effects of Glucagon-like peptide-1 (GLP-1) in the control of different cardiovascular pathologies and other effects beyond glycemic control, such as high blood pressure, weight control, and lipid metabolism. In addition to effects that are tangible in clinical practice, drugs that affect GLP-1 have been shown to have anti-atherosclerotic effects, due to the control of VR factors, or direct effects at the endothelial level. GLP-1-mediated decreases in atherosclerosis biomarkers, e.g., B-type natriuretic peptide (BNP), plasminogen activator inhibitor (PAI-1) and C- reactive protein (PCR), among others, have been observed. One of the parameters studied to validate this improvement in the progression of atherosclerosis has been the improvement in the control of the thickness of the carotid intima, which has clear benefits; however, studies in other vascular beds, such as the coronary, are more limited in terms of both numbers of participants and results.

The effect of semaglutide, a GLP-1 agonist, on the progression of atheroma plaque lesions has been published. Studies in animal models have shown that semaglutide treatment reduced progression by anti-inflammatory mechanisms, independent of weight loss and glycemic control. Semaglutide treatment in SUSTAIN6, as well as liraglutide treatment in LEADER, showed a benefit against placebo in major adverse cardiac events (MACE) (HR [95% confidence interval (CI)]: 0.87 [0.78; 0.97] LEADER and 0.74 [0.58; 0.95] SUSTAIN 6) in patients with atherosclerotic disease with or without previous ischemic events. The authors can affirm, after reviewing the literature, that the effect of GLP-1 on atheroma plaque is not definitively known but instead speculated on based on results in animal models and derived, to a large extent, from cardiovascular findings in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥35 and ≤ 65 years
* Absence of previous history of clinical cardiovascular events
* Subjects already taking therapy for diabetes on stable doses for 3 months or more.
* Subjects must have HbA1c at the initial screening visit between 8 and 10%
* Coronary CT performed less than 3 months before starting study medication

Exclusion Criteria:

* Clinically significant heart disease
* New York Heart Association (NYHA) class >II
* Known stroke or transient ischemic accident
* Uncontrolled hypertension at randomization, defined as a resting systolic blood pressure of 180 mm Hg at rest
* Personal or family history of hereditary muscular disorders
* Fasting triglyceride level > 250 mg/dL at screening
* Type 1 diabetes
* Known thyroid disease or subject taking thyroid replacement therapy
* Estimated glomerular filtration rate < 60 ml/min/1.73m2
* History of malignancy
* Known major active infection, or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction
* Baseline coronary CT does not meet Core Lab technical standards
* Cardiac rhythm different to normal sinus rhythm.
* Female subjects cannot be pregnant or breastfeeding, planning to become pregnant or planning to breastfeed during the entire study
* Premenopausal females of childbearing potential must be willing to use an acceptable method(s) of birth control during treatment and for an additional 15 weeks after the end of treatment

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plaque burden modification assessed by coronary CT and plaque quantification | 18 months
  The main objective of this trial is to evaluate the effect of Semaglutide on the burden of coronary atherosclerosis, based on the change in Percent Atheroma Volume (PAV) by quantifying atheroma plaque throughout the coronary tree based on the analysis of CCTA in asymptomatic subjects with T2D in optimized and stable treatment with Semaglutide

SECONDARY OUTCOMES:
Atheroma volume modification assessed by coronary CT and plaque quantification | 18 months
  Evaluate the effect of Semaglutide on the change in normalized total atheroma volume
Percentage of patients with significant plaque regresion assessed by coronary CT | 10 months
  Percentage of patients who demonstrated significant plaque regression
Changes in composition of artery wall assessed by coronary CT and plaque quantification | 18 months
  Effect of Semaglutide on the composition and architecture of the coronary artery wall
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 18 months
  Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Incidence of cardiovascular events | 18 months
  Incidence and type of cardiovascular events (cardiovascular death, Acute coronary syndrome and stroke) during treatment with Semaglutide.

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Pérez de Isla, Study Director — Hospital Clínico San Carlos. Madrid. Spain.

IPD SHARING:
Plan to Share IPD: Undecided